CLINICAL TRIAL: NCT05455255
Title: Application of the Web Program Based on the Flipped Model in Nursıng Process Teaching and Evaluation of Its Reflect to the Clinic
Brief Title: The Application of the Flipped Model in the Nursing Process and Evaluation of Its Reflection in the Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, nesibeyagmur, RESEARCH ASSISTANT, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20/01/2020-E.889
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Nursing Caries; Educational Problems
Keywords: Flipped Model; Nursing Process; Problem solving; Critical thinking

STUDY DESIGN:
Intervention Model Description: This research was planned to examine the effect of flipped learning on students' problem solving and critical thinking skills in nursing process teaching and their views on this model. In the quantitative part of this research, pretest-posttest randomized controlled experimental design, and in the qualitative part case study and phenomenological design will be used.
  Intervention and control groups will be determined by stratified randomization in line with the pre-test. In the quantitative design, flipped learning will be applied to the intervention group, while the traditional method will be applied to the control group. A focus group discussion will be held with the intervention group after the post-tests are administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): FL will be applied to the intervention group. In this model, short videos of the course will be delivered to students via WhatsApp one week in advance. At the beginning of the lesson, students' deficiencies will be corrected by making kahoot. Afterwards, group work, case scenario, role-play scenario and conceptual map methods will be applied in the course.
  Interventions: Other: Experimental
- Control Group (No Intervention): The subject of the nursing process will be transferred to the control group with powerpoint presentations by the educator. The activities in the other group will be presented by the trainer as an example.

INTERVENTIONS:
Other: Experimental — FL was applied by Jonathan Bergmann and Aaron Sams in 2007 for high school students who had to be absent from chemistry class. Bergmann and Sams published all the learning activities they used during the lesson as videos. Bergmann and Sams (2012) stated that in this model, which they developed over time, it is not compulsory for the trainer to explain the entire course content in the videos, and the important thing is to allocate time to active learning methods during the course. In the FL model, the summary of the course content is presented to the individuals outside the classroom with tools such as video and power point presentations. In the lesson, activities are carried out for the active participation of the student. The student performs the course content outside of the classroom, and the homework and learning the course in the classroom.
  Arms: Experimental Group

SUMMARY:
Teaching the nursing process that nursing students will use throughout their professional career is very important. In this direction, considering the Z generation, innovative and technology-based teaching methods should be used. Since the subject of the nursing process is the building block of nursing, its teaching should also be effective. The use of innovative and technology-based education methods that will increase the active participation of the students in the teaching of the nursing process, reinforce the learning, and encourage them to use problem-solving and critical thinking skills has been very important in recent years. For this reason, this research was planned to examine the effect of flipped learning(FL) on students' problem solving and critical thinking skills and their views on this model in nursing process teaching. In this study, it will be carried out with mixed method. In the quantitative part of the research, pre-test-post-test, experimental design with randomized control group will be used, and in the qualitative part, case study and phenomenological design will be used.

DETAILED DESCRIPTION:
Ethics committee approval was obtained from the Sakarya University Faculty of Medicine.In this study, it will be carried out with mixed method.

In the quantitative part of this research, pre-test-post-test, experimental design with randomized control group will be used, and in the qualitative part, case study and phenomenological design will be applied. Considering the losses as a result of the G-power analysis, the sample of the research was planned to consist of 23 students in the intervention group and 23 students in the control group. A stratified randomization process will be carried out by applying the pre-test data to the students who meet the inclusion criteria of the study.

In this study, FL will be applied to the intervention group for 5 weeks, while the traditional method will be applied to the control group for 5 weeks.

In the quantitative dimension of the research, critical thinking disposition scale and problem solving inventory will be used. A semi-structured interview form will be used in the qualitative aspect of the research.

ELIGIBILITY:
Inclusion Criteria:

Not having seen the subject of the nursing process before

* Adequate internet access
* Being willing to participate in the study.

Exclusion Criteria:

* Not willing to participate in the study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The genders were equalized in the experimental and control groups.
Enrollment: 46 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Critical Thinking Tendency Scale (CTTS) | 5 weeks
  In this study, the "Critical Thinking Tendency Scale (CTTS)" developed by Semerci (2016) was used. The Cronbach's alpha internal consistency coefficient of the CTTS scale was determined as 0.96. This scale consists of 49 items scaled as "I totally disagree (1)", I mostly disagree (2), I partially agree (3), I mostly agree (4), I totally agree (5)". The CTTS total score ranges from 49 to 245. It was stated that the students who scored high on the scale had a high tendency to think critically. (Semerci 2016).

SECONDARY OUTCOMES:
Problem Solving Inventory (PSI) | 5 weeks
  The Problem Solving Inventory used in the research is one of the tools that measures the individual's own perception of problem solving skills. The Cronbach's alpha internal consistency coefficient of the PSI scale was determined as 0.88. The Turkish adaptation of the scale developed by Heppner and Petersen in 1982 was carried out by Şahin, Şahin and Heppner (1993). A high total score from the scale indicates that individuals perceive themselves as inadequate in problem solving, while a low total score indicates that individuals perceive themselves as sufficient in problem solving skills

OTHER OUTCOMES:
Focus group semi-structured interview form -qualitative part | immediately after the intervention
  Semi-structured focus group interview forms were used in the qualitative part of this study, which was conducted with a mixed research design. Focus group interview forms contain open-ended questions and allow new questions to be added when there is a need to deepen on a topic during the interview. Interview questions were prepared by the researcher as a result of the literature review. Afterwards, opinions were taken by two different experts, and necessary adjustments were made in the focus group interview form in line with these opinions. The final version of the interview form consists of six open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Sakarya University, Principal Investigator — Sakarya University
Locations (1):
- Nasibe Yağmur Ziyai, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi H, Kim J, Bang KS, Park YH, Lee NJ, Kim C. Applying the Flipped Learning Model to an English-Medium Nursing Course. J Korean Acad Nurs. 2015 Dec;45(6):939-48. doi: 10.4040/jkan.2015.45.6.939. PMID 26805506
- [Result] Oh J, Kim SJ, Kim S, Kang KA, Kan J, Bartlett R. Development and evaluation of flipped learning using film clips within a nursing informatics course. Jpn J Nurs Sci. 2019 Oct;16(4):385-395. doi: 10.1111/jjns.12245. Epub 2018 Dec 19. PMID 30569630
- [Result] Kim Y, Kim N, Chae M. Effects of flipped learning on nursing students: A mixed methods study. Jpn J Nurs Sci. 2021 May 17:e12425. doi: 10.1111/jjns.12425. Online ahead of print. PMID 34002486
- [Result] Wassinger CA, Owens B, Boynewicz K, Williams DA. Flipped classroom versus traditional teaching methods within musculoskeletal physical therapy: a case report. Physiother Theory Pract. 2022 Nov;38(13):3169-3179. doi: 10.1080/09593985.2021.1941457. Epub 2021 Jun 28. PMID 34180751
- [Result] Njie-Carr VP, Ludeman E, Lee MC, Dordunoo D, Trocky NM, Jenkins LS. An Integrative Review of Flipped Classroom Teaching Models in Nursing Education. J Prof Nurs. 2017 Mar-Apr;33(2):133-144. doi: 10.1016/j.profnurs.2016.07.001. Epub 2016 Jul 22. PMID 28363388